CLINICAL TRIAL: NCT04117165
Title: Assessment of the Clinical and Medico-economic Impact of SinnoTest®, a Software That Predicts the Effectiveness of Biotherapy Treatments, in Patients With Rheumatoid Arthritis (RA)
Brief Title: Assessment of the Clinical and Medico-economic Impact of SinnoTest® in Patients With Rheumatoid Arthritis
Acronym: SINNO-RA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-A01709-48
Record Dates: First submitted 2019-09-30; First posted 2019-10-07 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Arthritis, Rheumatoid; Biological Therapy
Keywords: predictive software; quality of life
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Prospective clinical trial, phase III, randomized in 2 parallel groups, multicentric, controlled (prescription with SinnoTest® software versus prescription without SinnoTest® software), single-blind
Who Masked: Participant
Masking Description: The patient will not know if his bDMARD treatment was prescribed with or without the help of SinnoTest® software
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SinnoTest® software (Experimental): SinnoTest® is a therapeutic guidance device for patients suffering from chronic inflammatory rheumatism, in particular, rheumatoid arthritis. Prescription of bDMARD or their biosimilars is possible.
  Interventions: Diagnostic Test: Biotherapy Prescription with SinnoTest® software
- Patient Current care (Active Comparator): Current care of patients with rheumatoid arthritis, based on the recommendations of the French Society of Rheumatology. Prescription of bDMARD or their biosimilars is possible.
  Interventions: Drug: Patient Current Care

INTERVENTIONS:
Diagnostic Test: Biotherapy Prescription with SinnoTest® software — The rheumatologist will use the SinnoTest® software to give the best biotherapy to the patient according to the results of the software.
  Arms: SinnoTest® software
Drug: Patient Current Care — The rheumatologist will use the french guidelines of rheumatoid arthritis to choose the more adapted biotherapy treatment to the patient.
  Other Names: Biotherapy treatment without SinnoTest®
  Arms: Patient Current care

SUMMARY:
Rheumatoid arthritis (RA) is one of the main chronic inflammatory rheumatic diseases (RCI), with a prevalence of about 0.4% of the population.

First-line treatment with immunomodulators (synthetic and biological Disease Modifying Anti-Rheumatic Drugs (sDMARDs) including methotrexate) is not sufficiently effective in 40% of cases. These patients are then treated with biological Disease Modifying Anti-Rheumatic Drugs (bDMARDs) called biotherapies. As the use of these bio-drugs increases each year, they become a major public health and economic issue. Their growth is only just beginning, as they are among the major providers of pharmaceutical innovation.

There are about ten bio-drugs currently on the market for rheumatoid arthritis with an average annual treatment cost of 8 to 12 000 euros per patient. This cost is 20 times higher than that of sDMARDs. However, among patients treated with biotherapy, clinical practice shows that approximately one-third (33%) will not respond to the selected bio-drugs.

In the event of non-response, physicians currently have no choice but to rotate empirically between different treatments, as no tools capable of predicting response or non-response to these molecules are currently available. SinnoTest® software, a predictive algorithm for responding to bDMARDs by analyzing proteomic biomarkers, will clarify this choice of prescription for patients with failed RA of a first bDMARD in the anti-TNF family.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Rheumatoid Arthritis defined according to ACR/EULAR 2010 or ACR 1987 criteria.
* Patients in failure (patient insufficiently responding to anti-TNF treatment DAS28 > 3.2 whether related to primary biotherapy failure, loss of efficacy (loss of response) or adverse event) of a first bDMARD of the anti-TNF family (Adalimumab, Infliximab, Etanercept, Certolizumab or Golimumab).
* Stability of synthetic fund processing for 3 months.
* Corticosteroids ≤ 0.1 mg/kg/day without cortisone assault within 3 months.
* Effective contraception for patients with reproductive capacity (oral contraceptive, intrauterine device, implant, surgical sterilization or abstinence).
* Patients who have dated and signed the consent form for the trial.
* Patients affiliated to a social security system.

Exclusion Criteria:

* Contraindication to at least one of the following bDMARDs: Rituximab and/or Abatacept and/or Adalimumab.
* Scheduled surgical intervention during the trial.
* Difficulties in understanding the French language.
* Cognitive function disorders (dementia such as Alzheimer's, etc.).
* Patients who cannot be followed up at 12 months.
* Psycho-social instability incompatible with regular follow-up (homelessness, addictive behavior, a history of psychiatric pathology or any other comorbidity that would make free and informed consent impossible or limit adherence to the protocol).
* Persons referred to in Articles L1121-5 to L1121-8 of the CSP (corresponding to all protected persons: pregnant woman, parturient, breastfeeding mother, persons deprived of liberty by judicial or administrative decision, persons subject to a legal protection measure).
* Patients currently participating in other clinical research or who participated in a clinical trial within one month prior to inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit of using SinnoTest® software at 6 months | 6 months
  Clinical benefit of using SinnoTest® software in patients with RA who have failed to respond to a bDMARD of the anti-TNF family compared to usual care practice

SECONDARY OUTCOMES:
Clinical benefit of using SinnoTest® software at 1 year | 1 year
  Patients who respond according to the disease activity criteria from the DAS28 scale
Comparison of the response delay to a bDMARD and the number of bDMARDs prescribed during 12 months in both arms. | 1 year
  The delay and the number of bDMARDs prescribed before a good response
Performance of the software predictive model on the new clinical data from the trial at 6 months and 1 year | 6 months and 1 year
  Description of the properties of the prediction algorithms on the data of the study
Comparison of the variation in the proteomic profile between M0 (biotherapy start date) and M6 | Inclusion and 6 months
  Determination of the blood proteomic profile
Cost-utility analysis that will compare the 2 groups at 1 year from the community's perspective. | 1 year
  EuroQol five Dimensions questionnaire (EQ-5D-5L). The ratio will therefore be expressed as a cost per QALY earned, which represents the additional cost that will be required to earn a healthy year of life
Cost-effectiveness analysis that will compare the group with SinnoTest® compared to the group without SinnoTest®, at 1 year from the community's point of view. | 1 year
  Incremental Cost-Effectiveness Ratio (ICER)
Budget impact analysis from the point of view of Health Insurance at 3 and 5 years. | 3 and 5 years
  Measurement of the financial consequences for the Health Insurance of the implementation of SinnoTest® in the context of rheumatoid arthritis at 3- and 5-years' time point.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GAUDIN, PhD, Principal Investigator — University Hospital, Grenoble
Locations (16):
- France (16):
  - Chu Amiens, Amiens
  - CHU J Minjoz, Besançon
  - Groupe Hospitalier Pellegrin - CHU de Bordeaux, Bordeaux
  - CHU Cavale Blanche, Brest
  - Clinique de l'infirmerie protestante, Caluire-et-Cuire
  - Hôpital G. Montpied, Clermont-Ferrand
  - CHU DIJON Hôpital le Bocage, Dijon
  - Grenoble University Hospital, Grenoble
  - CHU Montpellier Hôpital Lapeyronie, Montpellier
  - CHU NANTES - Hôtel Dieu, Nantes
  - APHP Groupe hospitalier Pitié-Salpêtrière, Paris
  - APHP Hôpital Cochin, Paris
  - CHU Rouen Hôpital bois-guillaume, Rouen
  - CHU Saint-Etienne, Saint-Etienne
  - CHU Strasbourg Hôpital HAUTEPIERRE, Strasbourg
  - Hôpital PURPAN, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen MVC, Baillet A, Romand X, Trocme C, Courtier A, Marotte H, Thomas T, Soubrier M, Miossec P, Tebib J, Grange L, Toussaint B, Lequerre T, Vittecoq O, Gaudin P. Prealbumin, platelet factor 4 and S100A12 combination at baseline predicts good response to TNF alpha inhibitors in rheumatoid arthritis. Joint Bone Spine. 2019 Mar;86(2):195-201. doi: 10.1016/j.jbspin.2018.05.006. Epub 2018 Jun 6. PMID 29885551
- [Background] Nguyen MVC, Adrait A, Baillet A, Trocme C, Gottenberg JE, Gaudin P. Identification of cartilage oligomeric matrix protein as biomarker predicting abatacept response in rheumatoid arthritis patients with insufficient response to a first anti-TNFalpha treatment. Joint Bone Spine. 2019 May;86(3):401-403. doi: 10.1016/j.jbspin.2018.09.005. Epub 2018 Sep 19. No abstract available. PMID 30243783
- [Background] Baillet A, Trocme C, Romand X, Nguyen CMV, Courtier A, Toussaint B, Gaudin P, Epaulard O. Calprotectin discriminates septic arthritis from pseudogout and rheumatoid arthritis. Rheumatology (Oxford). 2019 Sep 1;58(9):1644-1648. doi: 10.1093/rheumatology/kez098. PMID 30919904
- [Background] Baillet A, Trocme C, Berthier S, Arlotto M, Grange L, Chenau J, Quetant S, Seve M, Berger F, Juvin R, Morel F, Gaudin P. Synovial fluid proteomic fingerprint: S100A8, S100A9 and S100A12 proteins discriminate rheumatoid arthritis from other inflammatory joint diseases. Rheumatology (Oxford). 2010 Apr;49(4):671-82. doi: 10.1093/rheumatology/kep452. Epub 2010 Jan 25. PMID 20100792
- [Background] Trocme C, Marotte H, Baillet A, Pallot-Prades B, Garin J, Grange L, Miossec P, Tebib J, Berger F, Nissen MJ, Juvin R, Morel F, Gaudin P. Apolipoprotein A-I and platelet factor 4 are biomarkers for infliximab response in rheumatoid arthritis. Ann Rheum Dis. 2009 Aug;68(8):1328-33. doi: 10.1136/ard.2008.093153. Epub 2008 Jul 29. PMID 18664547